CLINICAL TRIAL: NCT00069407
Title: Comparing Three Electrode Placements to Optimize ECT
Brief Title: Comparison of Three Electroconvulsive Therapy (ECT) Techniques for the Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH067201 (NIH); R01MH067201 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2003-09-24; First posted 2003-09-25 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: Bipolar Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RUL (Active Comparator): Right unilateral electroconvulsive therapy
  Interventions: Procedure: Electroconvulsive Therapy
- BL (Active Comparator): Bilateral electroconvulsive therapy
  Interventions: Procedure: Electroconvulsive Therapy
- BF (Active Comparator): Bifrontal electroconvulsive therapy
  Interventions: Procedure: Electroconvulsive Therapy

INTERVENTIONS:
Procedure: Electroconvulsive Therapy — Electroconvulsive therapy

SUMMARY:
This study will compare the antidepressant benefits and cognitive side effects of three different types of electroconvulsive therapy (ECT) in people with unipolar or bipolar depression.

DETAILED DESCRIPTION:
ECT is an important treatment for severely depressed people who do not respond adequately to, or are intolerant of, antidepressant medication. Traditionally, ECT has been administered with one of two standard techniques: bilateral and right unilateral electrode placement. However, these techniques are limited by either low efficacy or high cognitive impairment. Recently, an additional technique for ECT administration has shown promise in preliminary studies: bifrontal ECT. This study will compare this technique to the two traditional ECT techniques in treating people with depressive symptoms.

Participants in this study will be randomly assigned to receive standard bilateral ECT, high-dose right unilateral ECT, or bifrontal ECT in their index course. Depression symptoms, neuropsychological status, and quality of life will be measured throughout the course of the ECT treatment, one week after, and at a 2-month follow-up visit. This study will run for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar or bipolar depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2003-02; Primary Completion 2006-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, 24 item | 4 weeks
  Depression symptom rating

SECONDARY OUTCOMES:
Neuropsychological assessment | 4 weeks
  neuropsychological test battery

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Kellner, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - UMDNJ, Newark, New Jersey
  - Northshore/Long Island Jewish Hillside Hospital, Glen Oaks, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Kellner CH, Knapp R, Husain MM, Rasmussen K, Sampson S, Cullum M, McClintock SM, Tobias KG, Martino C, Mueller M, Bailine SH, Fink M, Petrides G. Bifrontal, bitemporal and right unilateral electrode placement in ECT: randomised trial. Br J Psychiatry. 2010 Mar;196(3):226-34. doi: 10.1192/bjp.bp.109.066183. PMID 20194546
- [Derived] Bailine S, Fink M, Knapp R, Petrides G, Husain MM, Rasmussen K, Sampson S, Mueller M, McClintock SM, Tobias KG, Kellner CH. Electroconvulsive therapy is equally effective in unipolar and bipolar depression. Acta Psychiatr Scand. 2010 Jun;121(6):431-6. doi: 10.1111/j.1600-0447.2009.01493.x. Epub 2009 Nov 8. PMID 19895623